CLINICAL TRIAL: NCT03334539
Title: A Phase 2, Multicenter, Randomized, Double-Masked and Placebo-Controlled Study Evaluating the Efficacy of Two Concentrations (0.10%, 0.25%) of HL036 Ophthalmic Solution Compared to Placebo in Subjects With Dry Eye
Brief Title: A Study to Assess Efficacy of HL036 in Subjects With Dry Eyes
Acronym: VELOS-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HanAll BioPharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HL036-DED-US-P201
Record Dates: First submitted 2017-10-11; First posted 2017-11-07 (Actual); Results first posted 2022-01-26 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2021-12

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 0.10% HL036 Ophthalmic Solution (Experimental): Participants self-administered HL036 0.10 percent (%) ophthalmic solution as topical ophthalmic drops, twice daily (BID) for up to 8 weeks. Exposures to the controlled adverse environment® (CAE) were conducted at Day 1, Day 15, Day 29 and Day 57.
  Interventions: Biological: HL036 ophthalmic solution
- 0.25% HL036 Ophthalmic Solution (Experimental): Participants self-administered HL036 0.25% ophthalmic solution as topical ophthalmic drops, BID for up to 8 weeks. Exposures to the CAE® were conducted at Day 1, Day 15, Day 29 and Day 57.
  Interventions: Biological: HL036 ophthalmic solution
- Placebo (Placebo Comparator): Participants self-administered HL036 placebo (vehicle solution) as topical ophthalmic drops, BID for up to 8 weeks. Exposures to the CAE® were conducted at Day 1, Day 15, Day 29 and Day 57.
  Interventions: Other: Placebo vehicle solution

INTERVENTIONS:
Biological: HL036 ophthalmic solution — HL036 ophthalmic solution
  Other Names: Tanfanercept
  Arms: 0.10% HL036 Ophthalmic Solution; 0.25% HL036 Ophthalmic Solution
Other: Placebo vehicle solution — Placebo vehicle solution
  Arms: Placebo

SUMMARY:
The objective of this study was to compare the safety and efficacy of 0.10% and 0.25% HL036 Ophthalmic Solutions to placebo for the treatment of the signs and symptoms of dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Have a patient-reported history of dry eye for at least 6 months prior to enrollment
* Have a history of use or desire to use eye drops for dry eye symptoms within 6 months of Visit 1
* Have in the study eye a Schirmer's Test score of ≤ 10 mm and ≥ 1 mm at Visits 1 and 2

Exclusion Criteria:

* Be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation at Visit 1
* Have used Restasis® or Xiidra® within 60 days of Visit 1
* Be currently taking any topical ophthalmic prescription (including medications for glaucoma) or over-the-counter (OTC) solutions, artificial tears, gels or scrubs, and cannot discontinue these medications for the duration of the trial (excluding medications allowed for the conduct of the study)
* Have an uncontrolled systemic disease
* Be a woman who is pregnant, nursing or planning a pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-11-05 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Torkildsen, MD, Principal Investigator — Andover Eye Associates
Locations (2):
- United States (2):
  - Central Maine Eye Care, Lewiston, Maine
  - Andover Eye Associates, Andover, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who met all the eligibility criteria were enrolled at 2 sites in the United States.
Pre-assignment Details: All participants went through a placebo run-in period for 14 days prior to randomization. During the period, exposures to the controlled adverse environment® (CAE) were conducted to ascertain eligibility to enter the study. Those who qualified were randomized.
Groups:
- 0.10% HL036 Ophthalmic Solution: Participants self-administered HL036 0.10 % ophthalmic solution as topical ophthalmic drops, twice daily (BID) for up to 8 weeks. Exposures to the controlled adverse environment (CAE®) were conducted at Day 1, Day 15, Day 29 and Day 57.
Period: Overall Study
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Started | 50 | 50 | 50
Completed | 46 | 43 | 49
Not Completed | 4 | 7 | 1
Not completed — Adverse Event | 3 | 5 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Administrative Reasons | 1 | 0 | 0
Not completed — Hypertension Not Controlled | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: The ITT population included all randomized participants.
Groups:
- 0.10% HL036 Ophthalmic Solution: Participants self-administered HL036 0.10 % ophthalmic solution as topical ophthalmic drops, BID for up to 8 weeks. Exposures to the CAE® were conducted at Day 1, Day 15, Day 29 and Day 57.
- Total: Total of all reporting groups
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo | Total
Number analyzed (Participants) | 50 | 50 | 50 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (13.09) | 63.5 (9.92) | 66.1 (11.38) | 63.5 (11.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 40 | 38 | 108
  Male | 20 | 10 | 12 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 2 | 5
  Not Hispanic or Latino | 48 | 49 | 48 | 145
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 49 | 48 | 48 | 145
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Coprimary Endpoint: Change From Baseline in Inferior Corneal Staining Score to Day 57 (Pre-CAE)
Description: It was evaluated for the inferior region on the Ora Calibra® Corneal and Conjunctival staining scale. The score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement.
Time Frame: Baseline (Day 1 Pre-CAE), Day 57 (Pre-CAE)
Population: ITT Population with the Markov Chain Monte Carlo (MCMC) imputation method for missing values.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: Participants self-administered HL036 placebo matching vehicle solution as topical ophthalmic drops, BID for up to 8 weeks. Exposures to the CAE® were conducted at Day 1, Day 15, Day 29 and Day 57.
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
score on a scale
  Day 1 Pre-CAE | 1.94 (0.512) | 1.96 (0.450) | 1.95 (0.433)
  Change From Baseline to Day 57 (pre-CAE) | 0.10 (0.699) | 0.10 (0.490) | -0.02 (0.631)
Statistical Analysis 1: Comparison: 0.10% HL036 Ophthalmic Solution vs Placebo; Test type: Superiority; p = 0.3378, ANCOVA — P-value was calculated using a model with treatment, baseline score, and site as covariates; Least Squares (LS) Mean Difference = 0.11, 95% CI 2-sided [-0.12 to 0.34]
Statistical Analysis 2: Comparison: 0.25% HL036 Ophthalmic Solution vs Placebo; Test type: Superiority; p = 0.2883, ANCOVA — P-value was calculated using a model with treatment, baseline score, and site as covariates; LS Mean Difference = 0.12, 95% CI 2-sided [-0.10 to 0.35]
Statistical Analysis 3: Comparison: 0.10% HL036 Ophthalmic Solution vs 0.25% HL036 Ophthalmic Solution; Test type: Other; p = 0.9293, ANCOVA — P-value calculated using a model with treatment, baseline score, and site as covariates; LS Mean Difference = 0.01, 95% CI 2-sided [-0.22 to 0.24]

2. Primary Outcome: Coprimary Endpoint: Change From Baseline in Ocular Discomfort Score to Day 57 (Pre-CAE)
Description: It is assessed by the Ora Calibra® Ocular Discomfort scale. The score ranged from 0 to 4 (0=none and 4=severe) with 1 point increments, where lower scores indicate improvement.
Time Frame: Baseline (Day 1 Pre-CAE), Day 57 (Pre-CAE)
Population: ITT Population with the MCMC imputation method for missing values.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
score on a scale
  Day 1 Pre-CAE | 2.6 (0.86) | 2.5 (0.95) | 2.4 (0.75)
  Change from Baseline: Day 57 (Pre-CAE) | -0.5 (1.16) | -0.4 (1.33) | -0.1 (0.88)
Statistical Analysis 1: Comparison: 0.10% HL036 Ophthalmic Solution vs Placebo; Test type: Superiority; p = 0.1473, ANCOVA — P-value calculated using a model with treatment, baseline score, and site as covariates; LS Mean Difference = -0.3, 95% CI 2-sided [-0.7 to 0.1]
Statistical Analysis 2: Comparison: 0.25% HL036 Ophthalmic Solution vs Placebo; Test type: Superiority; p = 0.2321, ANCOVA — P-value calculated using a model with treatment, baseline score, and site as covariates; LS Mean Difference = -0.3, 95% CI 2-sided [-0.7 to 0.2]
Statistical Analysis 3: Comparison: 0.10% HL036 Ophthalmic Solution vs 0.25% HL036 Ophthalmic Solution; Test type: Other; p = 0.8217, ANCOVA — P-value calculated using a model with treatment, baseline score, and site as covariates; LS Mean Difference = 0.0, 95% CI 2-sided [-0.4 to 0.5]

3. Secondary Outcome: Mean Change From Baseline in Fluorescein Staining (Inferior Region)
Description: It is evaluated for the inferior region on the Ora Calibra® Corneal and Conjunctival staining scale. The score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: Baseline (Day 1 Pre-CAE and Post-CAE), Day 8, Day 15 (Pre-CAE and Post-CAE), Day 29 (Pre-CAE and Post-CAE), and Day 57 (Pre-CAE and Post-CAE)
Population: Number of participants analyzed included participants in ITT Population with available data. The analysis was carried out with observed data only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
score on a scale
  Day 1 Pre-CAE | 1.94 (0.512) | 1.96 (0.450) | 1.95 (0.443)
  Day 1 Post-CAE | 3.32 (0.492) | 3.25 (0.565) | 3.20 (0.474)
  Day 1 (Change from Pre-CAE to Post-CAE) | 1.38 (0.521) | 1.29 (0.464) | 1.25 (0.407)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | 0.19 (0.706) | -0.01 (0.606) | 0.04 (0.668)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | -0.12 (0.697) | -0.20 (0.608) | -0.10 (0.571)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Post-CAE) | -0.62 (0.766) | -0.85 (0.736) | -0.69 (0.826)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.50 (0.892) | -0.66 (0.793) | -0.59 (0.867)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 29 (Pre-CAE) | 0.04 (0.807) | 0.04 (0.563) | 0.00 (0.707)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -0.41 (0.656) | -0.83 (0.677) | -0.48 (0.569)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.66 (0.857) | -1.02 (0.624) | -0.64 (0.591)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | 0.12 (0.724) | 0.10 (0.512) | -0.02 (0.631)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -0.47 (0.670) | -0.84 (0.738) | -0.63 (0.610)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.59 (0.878) | -0.92 (0.663) | -0.62 (0.747)

4. Secondary Outcome: Mean Change From Baseline in Fluorescein Staining (Superior Region)
Description: It is evaluated for the superior region on the Ora Calibra® Corneal and Conjunctival staining scale. The score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
score on a scale
  Day 1 Pre-CAE | 2.05 (0.420) | 2.08 (0.444) | 2.03 (0.456)
  Day 1 Post-CAE | 2.69 (0.552) | 2.56 (0.559) | 2.45 (0.556)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.64 (0.598) | 0.48 (0.622) | 0.42 (0.650)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | -0.09 (0.586) | -0.27 (0.592) | -0.09 (0.556)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | -0.22 (0.790) | -0.45 (0.724) | -0.29 (0.615)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Post-CAE) | -0.66 (0.976) | -0.72 (0.798) | -0.34 (0.658)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.44 (0.884) | -0.27 (0.743) | -0.05 (0.791)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 29 (Pre-CAE) | -0.27 (0.709) | -0.25 (0.555) | -0.10 (0.707)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -0.50 (0.655) | -0.65 (0.822) | -0.07 (0.604)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.41 (0.791) | -0.52 (0.964) | -0.09 (0.782)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | -0.09 (0.571) | -0.14 (0.594) | -0.19 (0.713)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -0.46 (0.665) | -0.37 (0.787) | -0.23 (0.662)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.37 (0.806) | -0.21 (0.847) | -0.08 (0.915)

5. Secondary Outcome: Mean Change From Baseline in Fluorescein Staining (Central Region)
Description: It is evaluated for the central region on the Ora Calibra® Corneal and Conjunctival staining scale. The score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
score on a scale
  Day 1 Pre-CAE | 1.45 (0.687) | 1.57 (0.670) | 1.49 (0.610)
  Day 1 Post-CAE | 2.22 (0.624) | 2.09 (0.550) | 2.04 (0.676)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.77 (0.641) | 0.052 (0.735) | 0.55 (0.633)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | 0.12 (0.766) | -0.02 (0.887) | -0.05 (0.779)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | 0.00 (0.869) | -0.24 (0.831) | -0.09 (0.780)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Post-CAE) | -0.52 (0.749) | -0.58 (0.732) | -0.42 (0.724)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.52 (0.963) | -0.34 (0.923) | -0.33 (0.956)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 29 (Pre-CAE) | 0.01 (0.906) | -0.21 (0.771) | -0.07 (0.776)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -0.50 (0.612) | -0.54 (0.528) | -0.16 (0.653)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.69 (0.870) | -0.54 (0.948) | -0.20 (0.916)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | 0.00 (0.837) | -0.10 (0.832) | -0.20 (0.802)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -0.36 (0.765) | -0.35 (0.856) | -0.30 (0.847)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.36 (1.089) | -0.23 (1.043) | -0.13 (0.846)

6. Secondary Outcome: Mean Change From Baseline in Fluorescein Staining (Temporal Region)
Description: It is evaluated for the temporal region on the Ora Calibra® Corneal and Conjunctival staining scale. The score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
score on a scale
  Day 1 Pre-CAE | 2.14 (0.452) | 2.12 (0.521) | 2.02 (0.622)
  Day 1 Post-CAE | 2.60 (0.606) | 2.42 (0.538) | 2.47 (0.519)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.46 (0.523) | 0.30 (0.647) | 0.45 (0.625)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | -0.01 (0.520) | -0.09 (0.598) | -0.13 (0.755)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | -0.34 (0.601) | -0.31 (0.741) | -0.14 (0.736)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Post-CAE) | -0.49 (0.739) | -0.54 (0.683) | -0.54 (0.552)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.15 (0.835) | -0.23 (0.765) | -0.40 (0.857)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 29 (Pre-CAE) | -0.19 (0.706) | -0.18 (0.828) | -0.10 (0.714)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -0.34 (0.569) | -0.38 (0.653) | -0.20 (0.478)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 27
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.26 (0.872) | -0.33 (0.894) | -0.20 (0.737)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | -0.07 (0.554) | 0.06 (0.749) | -0.09 (0.754)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -0.30 (0.679) | -0.24 (0.767) | -0.33 (0.696)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.24 (0.842) | -0.28 (0.902) | -0.26 (0.824)

7. Secondary Outcome: Mean Change From Baseline in Fluorescein Staining (Nasal Region)
Description: It is evaluated for the nasal region on the Ora Calibra® Corneal and Conjunctival staining scale. The score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
score on a scale
  Day 1 Pre-CAE | 2.27 (0.507) | 2.26 (0.527) | 2.14 (0.544)
  Day 1 Post-CAE | 2.74 (0.649) | 2.67 (0.577) | 2.68 (0.587)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.47 (0.557) | 0.41 (0.541) | 0.54 (0.638)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | -0.06 (0.501) | -0.05 (0.518) | -0.05 (0.702)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | -0.28 (0.743) | -0.29 (0.600) | -0.06 (0.620)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Post-CAE) | -0.44 (0.697) | -0.52 (0.785) | -0.51 (0.773)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.16 (0.830) | -0.23 (0.772) | -0.45 (0.859)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 29 (Pre-CAE) | -0.20 (0.735) | -0.18 (0.688) | -0.04 (0.783)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -0.17 (0.658) | -0.19 (0.694) | -0.20 (0.643)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 27
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.03 (0.755) | -0.06 (0.589) | -0.17 (0.877)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | -0.01 (0.771) | 0.01 (0.678) | -0.24 (0.600)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -0.29 (0.671) | -0.26 (0.960) | -0.38 (0.718)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.28 (0.696) | -0.27 (0.928) | -0.15 (0.805)

8. Secondary Outcome: Mean Change From Baseline in Fluorescein Staining (Corneal Sum)
Description: Corneal sum score is the sum of all regions of the cornea (inferior, superior and central regions). Individual region score was evaluated on the Ora Calibra® Corneal and Conjunctival staining scale. Individual region score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Corneal sum score ranges from 0 to 12. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
score on a scale
  Day 1 Pre-CAE | 5.44 (1.232) | 5.61 (1.230) | 5.47 (1.154)
  Day 1 Post-CAE | 8.23 (1.318) | 7.90 (1.241) | 7.69 (1.340)
  Day 1 (Change from Pre-CAE to Post-CAE) | 2.79 (1.258) | 2.29 (1.246) | 2.22 (1.135)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | 0.22 (1.559) | -0.30 (1.584) | -0.10 (1.544)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | -0.34 (1.939) | -0.89 (1.562) | -0.48 (1.474)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Post-CAE) | -1.80 (2.058) | -2.16 (1.695) | -1.45 (1.526)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -1.46 (1.935) | -1.27 (1.516) | -0.97 (1.739)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 29 (Pre-CAE) | -0.22 (1.995) | -0.42 (1.404) | -0.17 (1.704)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -1.41 (1.389) | -2.02 (1.360) | -0.71 (1.205)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -1.76 (1.850) | -2.08 (1.659) | -0.93 (1.438)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | 0.03 (1.470) | -0.14 (1.579) | -0.41 (1.634)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -1.28 (1.618) | -1.56 (1.780) | -1.16 (1.748)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -1.32 (2.034) | -1.36 (1.881) | -0.84 (1.801)

9. Secondary Outcome: Mean Change From Baseline in Fluorescein Staining (Conjunctival Sum)
Description: Conjunctival sum score is the sum of all regions of the conjunctiva (temporal and nasal regions). Individual region score was evaluated on the Ora Calibra® Corneal and Conjunctival staining scale. Individual region score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Conjunctival sum score ranges from 0 to 8. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
score on a scale
  Day 1 Pre-CAE | 4.41 (0.879) | 4.38 (0.923) | 4.16 (1.052)
  Day 1 Post-CAE | 5.34 (1.118) | 5.09 (0.941) | 5.15 (0.981)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.93 (0.827) | 0.71 (0.964) | 0.99 (1.095)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | -0.07 (0.845) | -0.15 (0.875) | -0.18 (1.349)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | -0.62 (1.167) | -0.60 (1.158) | -0.20 (1.143)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Post-CAE) | -0.93 (1.212) | -1.06 (1.295) | -1.05 (1.135)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.31 (1.269) | -0.46 (1.258) | -0.85 (1.440)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 29 (Pre-CAE) | -0.39 (1.263) | -0.35 (1.360) | -0.14 (1.327)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -0.52 (0.986) | -0.58 (1.206) | -0.39 (0.927)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 27
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.29 (1.379) | -0.38 (1.219) | -0.37 (1.377)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | -0.08 (1.178) | 0.07 (1.269) | -0.33 (1.223)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -0.60 (1.177) | -0.50 (1.528) | -0.70 (1.194)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.52 (1.273) | -0.55 (1.573) | -0.41 (1.306)

10. Secondary Outcome: Mean Change From Baseline in Fluorescein Staining Total Score (All Five Regions: Central, Superior, Inferior, Temporal, Nasal)
Description: Total score was sum of all 5 regions: central, superior, inferior, temporal, and nasal. Individual region score was evaluated on the Ora Calibra® Corneal and Conjunctival staining scale. Individual region score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Total score ranges from 0 to 20. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
score on a scale
  Day 1 Pre-CAE | 9.85 (1.852) | 9.99 (1.777) | 9.63 (1.982)
  Day 1 Post-CAE | 13.57 (2.143) | 12.99 (1.828) | 12.84 (1.872)
  Day 1 (Change from Pre-CAE to Post-CAE) | 3.72 (1.614) | 3.00 (1.684) | 3.21 (1.890)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | 0.15 (2.139) | -0.45 (2.009) | -0.29 (2.667)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | -0.96 (2.866) | -1.49 (2.312) | -0.68 (2.338)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Post-CAE) | -2.73 (2.875) | -3.22 (2.664) | -2.50 (2.150)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -1.77 (2.686) | -1.73 (2.245) | -1.82 (2.676)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 29 (Pre-CAE) | -0.61 (2.933) | -0.77 (2.214) | -0.30 (2.710)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -1.93 (1.831) | -2.60 (2.168) | -1.11 (1.739)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 27
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -2.05 (2.530) | -2.46 (2.054) | -1.30 (2.403)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | -0.04 (2.250) | -0.07 (2.403) | -0.74 (2.560)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -1.88 (2.400) | -2.06 (2.990) | -1.87 (2.559)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -1.84 (2.763) | -1.91 (2.922) | -1.24 (2.387)

11. Secondary Outcome: Mean Change From Baseline in Lissamine Green Staining Total Score (Inferior Region)
Description: It is evaluated for the inferior region on the lissamine green corneal and conjunctival staining scale (Ora Calibra® scale). Individual region score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 0.10% HL036 Ophthalmic Solution: Participants self-administered HL036 0.10% ophthalmic solution as topical ophthalmic drops, BID for up to 8 weeks. Exposures to the CAE® were conducted at Day 1, Day 15, Day 29 and Day 57.
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
score on a scale
  Day 1 Pre-CAE | 1.42 (0.642) | 1.46 (0.605) | 1.50 (0.580)
  Day 1 Post-CAE | 2.00 (0.920) | 2.12 (0.895) | 1.87 (0.826)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.58 (0.752) | 0.66 (0.934) | 0.37 (0.850)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | 0.04 (0.699) | -0.30 (0.642) | -0.08 (0.702)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | -0.34 (0.805) | -0.43 (0.644) | -0.48 (0.707)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Post-CAE) | -0.46 (1.228) | -0.76 (0.984) | -0.34 (1.104)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.12 (0.982) | -0.33 (0.919) | 0.14 (1.170)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 29 (Pre-CAE) | -0.14 (0.815) | -0.24 (0.715) | -0.28 (0.607)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -0.10 (1.191) | -0.69 (0.895) | -0.20 (1.074)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.10 (1.064) | -0.60 (0.949) | 0.16 (1.147)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | -0.21 (0.637) | -0.17 (0.869) | -0.34 (0.688)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -0.16 (0.943) | -0.60 (0.877) | -0.22 (0.764)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | 0.04 (0.881) | -0.38 (1.179) | 0.07 (0.866)

12. Secondary Outcome: Mean Change From Baseline in Lissamine Green Staining Total Score (Superior Region)
Description: It is evaluated for the superior region on the lissamine green corneal and conjunctival staining scale (Ora Calibra® scale). Individual region score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
score on a scale
  Day 1 Pre-CAE | 1.22 (0.507) | 1.32 (0.560) | 1.27 (0.546)
  Day 1 Post-CAE | 1.48 (0.580) | 1.51 (0.703) | 1.44 (0.697)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.26 (0.527) | 0.19 (0.669) | 0.17 (0.760)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | -0.14 (0.525) | -0.31 (0.624) | -0.18 (0.537)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | -0.37 (0.838) | -0.57 (0.772) | -0.38 (0.907)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Post-CAE) | -0.48 (0.931) | -0.66 (0.870) | -0.34 (0.866)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.11 (0.841) | -0.08 (0.808) | 0.04 (0.936)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 29 (Pre-CAE) | -0.29 (0.729) | -0.33 (0.604) | -0.44 (0.712)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -0.19 (0.806) | -0.31 (0.849) | 0.02 (0.713)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.14 (0.789) | -0.04 (0.916) | 0.30 (0.896)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | -0.32 (0.541) | -0.36 (0.694) | -0.40 (0.769)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -0.37 (0.679) | -0.44 (0.717) | -0.28 (0.736)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.05 (0.797) | -0.05 (0.762) | 0.08 (0.915)

13. Secondary Outcome: Mean Change From Baseline in Lissamine Green Staining Total Score (Central Region)
Description: It is evaluated for the central region on the lissamine green corneal and conjunctival staining scale (Ora Calibra® scale). Individual region score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
score on a scale
  Day 1 Pre-CAE | 0.48 (0.735) | 0.57 (0.742) | 0.54 (0.734)
  Day 1 Post-CAE | 0.59 (0.780) | 0.60 (0.735) | 0.66 (0.823)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.11 (0.547) | 0.03 (0.519) | 0.12 (0.799)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | -0.13 (0.676) | -0.29 (0.582) | -0.24 (0.723)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | -0.13 (0.720) | -0.26 (0.636) | -0.24 (0.744)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Post-CAE) | -0.33 (0.636) | -0.29 (0.706) | -0.30 (0.647)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.20 (0.776) | -0.03 (0.815) | -0.06 (0.935)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 29 (Pre-CAE) | -0.31 (0.630) | -0.22 (0.837) | -0.28 (0.730)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -0.07 (0.258) | -0.15 (0.660) | -0.07 (0.466)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | 0.03 (0.680) | -0.17 (0.677) | 0.11 (0.956)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | -0.23 (0.555) | -0.31 (0.667) | -0.16 (0.681)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -0.14 (0.602) | -0.34 (0.898) | -0.31 (0.619)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | 0.09 (0.652) | -0.02 (0.879) | -0.18 (0.782)

14. Secondary Outcome: Mean Change From Baseline in Lissamine Green Staining Total Score (Temporal Region)
Description: It is evaluated for the temporal region on the lissamine green corneal and conjunctival staining scale (Ora Calibra® scale). Individual region score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
score on a scale
  Day 1 Pre-CAE | 1.63 (0.706) | 1.63 (0.669) | 1.61 (0.751)
  Day 1 Post-CAE | 1.87 (0.691) | 1.71 (0.671) | 1.87 (0.734)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.24 (0.649) | 0.08 (0.695) | 0.26 (0.834)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | -0.09 (0.733) | -0.11 (0.864) | -0.15 (0.686)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | -0.32 (0.885) | -0.48 (0.707) | -0.46 (0.885)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Post-CAE) | -0.37 (0.669) | -0.50 (0.772) | -0.50 (0.606)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.05 (0.876) | -0.02 (0.928) | -0.04 (0.919)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 29 (Pre-CAE) | -0.29 (0.915) | -0.21 (0.683) | -0.19 (0.630)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -0.28 (0.663) | -0.06 (0.668) | -0.25 (0.569)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.09 (1.142) | 0.08 (0.688) | -0.05 (0.916)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | -0.26 (0.721) | -0.20 (0.816) | -0.16 (0.710)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -0.21 (0.750) | -0.22 (0.934) | -0.22 (0.715)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | 0.05 (1.029) | 0.03 (0.947) | -0.07 (1.066)

15. Secondary Outcome: Mean Change From Baseline in Lissamine Green Staining Total Score (Nasal Region)
Description: It is evaluated for the nasal region on the lissamine green corneal and conjunctival staining scale (Ora Calibra® scale). Individual region score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
score on a scale
  Day 1 Pre-CAE | 1.90 (0.707) | 1.96 (0.561) | 1.69 (0.638)
  Day 1 Post-CAE | 2.18 (0.774) | 2.05 (0.828) | 1.93 (0.693)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.28 (0.640) | 0.09 (0.740) | 0.24 (0.816)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | -0.04 (0.748) | -0.25 (0.668) | 0.00 (0.677)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | -0.22 (0.723) | -0.48 (0.660) | -0.23 (0.822)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Post-CAE) | -0.23 (0.858) | -0.29 (0.904) | -0.24 (0.672)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.01 (0.901) | 0.19 (1.070) | -0.01 (1.013)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 29 (Pre-CAE) | -0.28 (0.679) | -0.39 (0.638) | -0.03 (0.785)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -0.19 (0.737) | 0.10 (0.749) | -0.11 (0.854)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | 0.09 (0.780) | 0.52 (0.781) | -0.02 (1.004)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | -0.12 (0.709) | -0.31 (0.692) | -0.10 (0.721)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -0.26 (0.815) | -0.16 (0.843) | -0.02 (0.841)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.14 (0.821) | 0.17 (0.872) | 0.05 (0.959)

16. Secondary Outcome: Mean Change From Baseline in Lissamine Green Staining Total Score (Corneal Sum)
Description: Corneal sum score is the sum of all regions of the cornea (inferior, superior and central regions). Individual region score was evaluated on the lissamine green corneal and conjunctival staining scale (Ora Calibra® scale). Individual region score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Total score ranges from 0 to 12. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
score on a scale
  Day 1 Pre-CAE | 3.12 (1.272) | 3.35 (1.360) | 3.31 (1.344)
  Day 1 Post-CAE | 4.07 (1.705) | 4.23 (1.785) | 3.97 (1.828)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.95 (1.314) | 0.88 (1.683) | 0.66 (1.701)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | -0.23 (1.258) | -0.91 (1.382) | -0.51 (1.375)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | -0.84 (1.633) | -1.26 (1.568) | -1.10 (1.909)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Post-CAE) | -1.27 (2.264) | -1.71 (2.118) | -0.98 (1.924)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.43 (1.648) | -0.45 (1.952) | 0.12 (1.965)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 29 (Pre-CAE) | -0.74 (1.516) | -0.79 (1.487) | -1.00 (1.488)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -0.36 (1.782) | -1.15 (1.754) | -0.25 (1.430)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.21 (1.578) | -0.81 (1.588) | 0.57 (1.783)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | -0.75 (1.228) | -0.84 (1.751) | -0.90 (1.793)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -0.67 (1.674) | -1.38 (1.936) | -0.81 (1.439)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | 0.08 (1.494) | -0.45 (2.154) | -0.03 (1.586)

17. Secondary Outcome: Mean Change From Baseline in Lissamine Green Staining Total Score (Conjunctival Sum)
Description: Conjunctival sum score is the sum of all regions of the conjunctiva (temporal and nasal regions). Individual region score was evaluated on the lissamine green corneal and conjunctival staining scale (Ora Calibra® scale). Individual region score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Total score ranges from 0 to 8. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
score on a scale
  Day 1 Pre-CAE | 3.53 (1.231) | 3.59 (1.058) | 3.30 (1.237)
  Day 1 Post-CAE | 4.05 (1.314) | 3.76 (1.322) | 3.80 (1.262)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.52 (1.092) | 0.17 (1.223) | 0.50 (1.403)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | -0.13 (1.249) | -0.36 (1.197) | -0.15 (1.133)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | -0.54 (1.417) | -0.96 (1.056) | -0.69 (1.548)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Post-CAE) | -0.60 (1.245) | -0.79 (1.228) | -0.74 (1.084)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.06 (1.427) | 0.17 (1.524) | -0.05 (1.724)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 29 (Pre-CAE) | -0.57 (1.336) | -0.59 (1.090) | -0.22 (1.112)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -0.47 (1.195) | 0.04 (1.264) | -0.36 (1.154)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | 0.00 (1.553) | 0.60 (1.200) | -0.07 (1.412)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | -0.38 (1.175) | -0.51 (1.349) | -0.26 (1.222)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -0.47 (1.356) | -0.38 (1.577) | -0.24 (1.377)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.09 (1.668) | 0.21 (1.461) | -0.02 (1.723)

18. Secondary Outcome: Mean Change From Baseline in Lissamine Green Staining Total Score (All Five Regions: Central, Superior, Inferior, Temporal, Nasal)
Description: Total score was sum of all 5 regions: central, superior, inferior, temporal, and nasal. Individual region score was evaluated on the lissamine green corneal and conjunctival staining scale (Ora Calibra® scale). Individual region score ranges from 0 to 4 (0=none and 4=severe), and lower score indicates improvement. Total score ranges from 0 to 20. Change score from pre- to post-CAE® was calculated as post-CAE® score - pre-CAE® score.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
score on a scale
  Day 1 Pre-CAE | 6.65 (2.277) | 6.94 (2.091) | 6.61 (2.223)
  Day 1 Post-CAE | 8.12 (2.653) | 7.99 (2.753) | 7.77 (2.741)
  Day 1 (Change from Pre-CAE to Post-CAE) | 1.47 (1.923) | 1.05 (2.493) | 1.16 (2.708)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | -0.36 (2.124) | -1.27 (2.065) | -0.66 (2.090)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | -1.38 (2.767) | -2.22 (2.193) | -1.79 (3.059)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Post-CAE) | -1.87 (3.156) | -2.50 (2.836) | -1.72 (2.607)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.49 (2.409) | -0.28 (2.633) | 0.07 (3.161)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 29 (Pre-CAE) | -1.31 (2.435) | -1.39 (2.038) | -1.22 (2.150)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -0.83 (2.369) | -1.12 (2.455) | -0.61 (2.025)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.21 (2.551) | -0.21 (2.016) | 0.50 (2.553)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | -1.13 (1.815) | -1.35 (2.684) | -1.16 (2.616)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -1.14 (2.635) | -1.77 (3.087) | -1.05 (2.424)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.01 (2.568) | -0.24 (3.138) | -0.05 (2.716)

19. Secondary Outcome: Change From Baseline in Tear Film Break-Up Time
Description: Sodium fluorescein solution was instilled into each eye and participants were instructed to blinked several times. The time it takes to form micelles from the time that the eye is opened was noted.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
seconds
  Day 1 Pre-CAE | 1.559 (0.5031) | 1.709 (0.7083) | 1.574 (0.5394)
  Day 1 Post-CAE | 1.533 (0.5217) | 1.555 (0.5441) | 1.574 (0.5322)
  Day 1 (Change from Pre-CAE to Post-CAE) | -0.027 (0.4552) | -0.154 (0.5516) | -0.001 (0.3670)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | 0.024 (0.4943) | -0.037 (0.7421) | -0.036 (0.4948)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | 0.386 (0.8008) | 0.127 (0.7945) | 0.276 (0.7857)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Post-CAE) | 0.312 (0.9470) | 0.195 (0.6835) | 0.222 (0.7884)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.075 (0.7355) | 0.068 (0.6543) | -0.054 (0.6252)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 29 (Pre-CAE) | 0.218 (0.7586) | -0.191 (0.5936) | -0.077 (0.5228)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | 0.123 (0.7116) | 0.086 (0.6752) | -0.188 (0.3884)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.054 (0.5013) | 0.129 (0.4258) | -0.119 (0.5623)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | 0.139 (0.5727) | -0.036 (0.8880) | 0.186 (0.6696)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | 0.118 (0.7072) | 0.039 (0.6057) | 0.160 (0.7206)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.021 (0.6113) | 0.063 (0.8557) | -0.003 (0.6473)

20. Secondary Outcome: Change From Baseline in the Ora Calibra® Conjunctival Redness Scale
Description: It is evaluated by the Ora Calibra® conjunctival redness scale for dry eye. The score ranges from 0 to 4 (0=none and 4=severe), where lower score indicates improvement
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
score on a scale
  Day 1 Pre-CAE | 1.70 (0.639) | 1.66 (0.566) | 1.72 (0.536)
  Day 1 Post-CAE | 2.03 (0.626) | 2.02 (0.571) | 2.04 (0.523)
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.33 (0.603) | 0.36 (0.655) | 0.32 (0.569)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | 0.04 (0.588) | -0.07 (0.473) | 0.00 (0.669)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | -0.20 (0.606) | -0.17 (0.559) | -0.17 (0.568)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Post-CAE) | -0.14 (0.663) | -0.35 (0.515) | -0.20 (0.606)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | 0.06 (0.983) | -0.19 (0.836) | -0.03 (0.785)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 29 (Pre-CAE) | -0.06 (0.740) | -0.03 (0.614) | -0.10 (0.685)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -0.22 (0.635) | -0.31 (0.601) | -0.21 (0.568)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.05 (0.967) | -0.21 (0.907) | -0.11 (1.012)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | 0.01 (0.563) | 0.23 (0.660) | 0.11 (0.565)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -0.03 (0.591) | -0.01 (0.728) | -0.14 (0.586)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.04 (0.788) | -0.22 (0.941) | -0.28 (0.708)

21. Secondary Outcome: Change From Baseline in Schirmer's Test
Description: The Schirmer test strip will be placed in the lower temporal lid margin of each eye. Subjects will be instructed to close their eyes and After 5 minutes have elapsed, The length of moistened area of schirmer strip will be recorded (mm) for each eye.
Time Frame: Baseline (Day 1); Days 15, 29, and 57
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Groups:
- 0.10% HL036 Ophthalmic Solution: Participants self-administered HL036 0.10 percent (%) ophthalmic solution as topical ophthalmic drops, twice daily (BID) for up to 8 weeks. Exposures to the controlled adverse environment® (CAE) were conducted at Day 15, Day 29 and Day 57.
- 0.25% HL036 Ophthalmic Solution: Participants self-administered HL036 0.25% ophthalmic solution as topical ophthalmic drops, BID for up to 8 weeks. Exposures to the controlled adverse environment® (CAE) were conducted at Day 15, Day 29 and Day 57.
- Placebo: Participants sefl-administered HL036 placebo matching vehicle solution as topical ophthalmic drops, BID for up to 8 weeks. Exposures to the controlled adverse environment® (CAE) were conducted at Day 15, Day 29 and Day 57.
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
mm
  Day 1 | 5.0 (2.60) | 5.2 (3.03) | 5.5 (3.02)
  Change From Baseline: Day 15: number analyzed (Participants) | 50 | 48 | 50
  Change From Baseline: Day 15 | 1.7 (5.21) | 4.0 (7.36) | 3.4 (6.50)
  Change From Baseline: Day 29: number analyzed (Participants) | 50 | 47 | 50
  Change From Baseline: Day 29 | 0.8 (5.01) | 0.9 (4.23) | 1.8 (4.35)
  Change From Baseline: Day 57: number analyzed (Participants) | 46 | 43 | 49
  Change From Baseline: Day 57 | 3.5 (6.70) | 2.9 (4.74) | 3.3 (6.84)

22. Secondary Outcome: Change From Baseline in Ora Calibra® Ocular Discomfort Scale
Description: It was assessed by the Ora Calibra® ocular discomfort scale. The score ranges from 0 to 4 (0=none and 4=severe), where lower score indicates improvement.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
score on a scale
  Day 1 Pre-CAE | 2.6 (0.86) | 2.5 (0.95) | 2.4 (0.75)
  Day 1 Post-CAE: number analyzed (Participants) | 50 | 49 | 50
  Day 1 Post-CAE | 3.8 (0.52) | 3.7 (0.47) | 3.8 (0.52)
  Day 1 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 49 | 50
  Day 1 (Change from Pre-CAE to Post-CAE) | 1.2 (0.98) | 1.2 (1.01) | 1.4 (0.81)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | -0.5 (0.89) | 0.1 (0.81) | -0.1 (1.01)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | -0.5 (0.71) | -0.1 (0.96) | -0.1 (0.87)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Post-CAE) | 0.0 (0.62) | 0.0 (0.58) | 0.0 (0.55)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | 0.5 (0.91) | 0.1 (1.13) | 0.1 (1.05)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 29 (Pre-CAE) | -0.4 (1.03) | -0.3 (0.92) | -0.2 (1.05)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | 0.0 (0.63) | -0.2 (0.63) | 0.0 (0.88)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | 0.5 (1.18) | 0.0 (1.11) | 0.1 (1.36)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | -0.5 (1.17) | -0.4 (1.39) | -0.1 (0.88)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -0.2 (0.77) | -0.1 (0.65) | -0.2 (0.76)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | 0.3 (1.30) | 0.4 (1.43) | -0.1 (1.17)

23. Secondary Outcome: Change From Baseline in Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire for Dry Eye (Overall Ocular Discomfort)
Description: Ora Calibra® ocular discomfort & 4-symptom questionnaire for dry eye includes rating of the severity of 5 symptoms: ocular discomfort, burning, dryness, grittiness, and stinging.
  Participants rated the severity of overall ocular discomfort at all scheduled visits on 0 to 5 scale, where 0=none and 5=severe. Higher score represent higher severity.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
score on a scale
  Day 1 Pre-CAE: number analyzed (Participants) | 50 | 50 | 48
  Day 1 Pre-CAE | 2.9 (0.88) | 2.7 (1.09) | 2.8 (0.78)
  Day 1 Post-CAE: number analyzed (Participants) | 50 | 49 | 50
  Day 1 Post-CAE | 3.8 (0.57) | 3.7 (0.81) | 4.0 (0.74)
  Day 1 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 49 | 48
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.9 (0.82) | 1.0 (1.11) | 1.2 (0.92)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | -0.3 (0.97) | 0.0 (0.98) | -0.2 (0.90)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | -0.4 (0.93) | 0.0 (1.00) | -0.1 (0.97)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 47 | 50
  Change from Baseline: Day 15 (Post-CAE) | -0.2 (0.78) | 0.0 (0.66) | -0.2 (0.95)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 47 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | 0.2 (1.13) | 0.0 (1.07) | 0.0 (1.40)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 29 (Pre-CAE) | -0.3 (1.05) | -0.3 (1.19) | -0.3 (1.17)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -0.1 (0.90) | 0.0 (0.89) | -0.1 (0.72)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | 0.3 (1.03) | 0.3 (1.23) | 0.2 (1.49)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | -0.5 (1.35) | -0.4 (1.35) | -0.2 (1.06)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -0.2 (0.86) | 0.0 (0.64) | -0.4 (0.98)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | 0.3 (1.47) | 0.5 (1.32) | -0.1 (1.33)

24. Secondary Outcome: Change From Baseline in Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire for Dry Eye (Burning)
Description: Ora Calibra® ocular discomfort & 4-symptom questionnaire for dry eye includes rating of the severity of 5 symptoms: ocular discomfort, burning, dryness, grittiness, and stinging.
  Participants rated the severity of burning at all scheduled visits on 0 to 5 scale, where 0=none and 5=severe. Higher score represent higher severity.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
score on a scale
  Day 1 Pre-CAE | 1.6 (1.31) | 1.4 (1.35) | 1.2 (1.28)
  Day 1 Post-CAE: number analyzed (Participants) | 50 | 49 | 50
  Day 1 Post-CAE | 2.5 (1.49) | 2.3 (1.55) | 2.4 (1.66)
  Day 1 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 49 | 50
  Day 1 (Change from Pre-CAE to Post-CAE) | 1.0 (1.26) | 0.9 (1.12) | 1.2 (1.29)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | -0.1 (0.81) | 0.0 (0.92) | 0.0 (0.85)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | -0.1 (1.04) | -0.2 (1.14) | 0.0 (0.74)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 47 | 50
  Change from Baseline: Day 15 (Post-CAE) | -0.1 (1.16) | 0.0 (1.17) | -0.1 (1.05)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 47 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | 0.0 (1.62) | 0.2 (1.40) | -0.1 (1.40)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 29 (Pre-CAE) | -0.1 (1.14) | -0.2 (1.18) | 0.0 (0.84)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -0.1 (1.35) | -0.2 (0.97) | -0.1 (0.85)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | 0.1 (1.25) | 0.4 (1.24) | -0.3 (1.21)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | -0.1 (1.22) | -0.5 (1.50) | -0.1 (0.93)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -0.2 (1.09) | -0.1 (1.28) | -0.3 (1.01)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.1 (1.48) | 0.5 (1.26) | -0.2 (1.30)

25. Secondary Outcome: Change From Baseline in Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire for Dry Eye (Dryness)
Description: Ora Calibra® ocular discomfort & 4-symptom questionnaire for dry eye includes rating of the severity of 5 symptoms: ocular discomfort, burning, dryness, grittiness, and stinging.
  Participants rated the severity of dryness at all scheduled visits on 0 to 5 scale, where 0=none and 5=severe. Higher score represent higher severity.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
score on a scale
  Day 1 Pre-CAE | 3.1 (0.87) | 3.1 (1.03) | 3.0 (0.84)
  Day 1 Post-CAE: number analyzed (Participants) | 50 | 49 | 50
  Day 1 Post-CAE | 4.0 (0.71) | 3.9 (0.80) | 4.1 (0.63)
  Day 1 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 49 | 50
  Day 1 (Change from Pre-CAE to Post-CAE) | 1.0 (0.86) | 0.9 (0.76) | 1.1 (0.99)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | -0.4 (0.90) | -0.1 (0.70) | -0.2 (0.77)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | -0.3 (0.80) | -0.2 (0.90) | -0.1 (0.76)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 47 | 50
  Change from Baseline: Day 15 (Post-CAE) | -0.2 (0.71) | -0.2 (0.80) | -0.1 (0.95)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 47 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | 0.1 (1.08) | 0.0 (0.98) | 0.0 (1.29)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 29 (Pre-CAE) | -0.2 (1.03) | -0.4 (1.01) | -0.3 (0.94)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -0.3 (1.04) | -0.2 (0.67) | -0.2 (0.79)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | 0.0 (0.98) | 0.5 (1.17) | 0.1 (1.33)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | -0.4 (1.25) | -0.3 (1.20) | -0.2 (1.08)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -0.2 (0.85) | -0.1 (0.82) | -0.3 (1.09)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | 0.1 (1.31) | 0.3 (1.04) | -0.1 (1.36)

26. Secondary Outcome: Change From Baseline in Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire for Dry Eye (Grittiness)
Description: Ora Calibra® ocular discomfort & 4-symptom questionnaire for dry eye includes rating of the severity of 5 symptoms: ocular discomfort, burning, dryness, grittiness, and stinging.
  Participants rated the severity of grittiness at all scheduled visits on 0 to 5 scale, where 0=none and 5=severe. Higher score represent higher severity.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
score on a scale
  Day 1 Pre-CAE | 2.1 (1.27) | 1.8 (1.47) | 2.0 (1.35)
  Day 1 Post-CAE: number analyzed (Participants) | 50 | 49 | 50
  Day 1 Post-CAE | 2.7 (1.40) | 2.3 (1.63) | 3.0 (1.28)
  Day 1 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 49 | 50
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.7 (1.10) | 0.5 (0.96) | 1.1 (1.10)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | -0.2 (1.06) | -0.1 (0.67) | 0.1 (0.95)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | -0.1 (1.05) | 0.2 (1.06) | 0.0 (0.68)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 47 | 50
  Change from Baseline: Day 15 (Post-CAE) | -0.1 (1.00) | 0.2 (1.24) | -0.3 (1.07)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 47 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | 0.0 (1.29) | 0.0 (1.03) | -0.3 (1.33)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 29 (Pre-CAE) | -0.2 (1.25) | -0.1 (1.18) | -0.2 (1.04)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -0.2 (0.99) | 0.1 (1.03) | -0.1 (0.74)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | 0.1 (1.18) | 0.3 (1.01) | 0.0 (1.22)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | -0.4 (1.20) | -0.1 (1.29) | -0.1 (0.94)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -0.3 (1.06) | 0.2 (1.13) | -0.6 (1.08)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | 0.0 (1.44) | 0.3 (1.09) | -0.4 (1.14)

27. Secondary Outcome: Change From Baseline in Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire for Dry Eye (Stinging)
Description: Ora Calibra® ocular discomfort & 4-symptom questionnaire for dry eye includes rating of the severity of 5 symptoms: ocular discomfort, burning, dryness, grittiness, and stinging.
  Participants rated the severity of stinging at all scheduled visits on 0 to 5 scale, where 0=none and 5=severe. Higher score represent higher severity.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
score on a scale
  Day 1 Pre-CAE | 1.5 (1.33) | 1.2 (1.35) | 1.0 (1.08)
  Day 1 Post-CAE: number analyzed (Participants) | 50 | 49 | 50
  Day 1 Post-CAE | 2.3 (1.42) | 1.9 (1.55) | 2.0 (1.67)
  Day 1 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 49 | 50
  Day 1 (Change from Pre-CAE to Post-CAE) | 0.8 (1.18) | 0.7 (1.05) | 1.0 (1.26)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | -0.3 (0.92) | -0.2 (0.86) | -0.1 (0.69)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | -0.2 (1.04) | -0.2 (1.08) | 0.0 (0.76)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 49 | 47 | 50
  Change from Baseline: Day 15 (Post-CAE) | -0.3 (1.12) | 0.0 (1.00) | -0.1 (1.19)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 49 | 47 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | 0.0 (1.34) | 0.2 (1.24) | -0.1 (1.41)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 29 (Pre-CAE) | -0.2 (1.12) | -0.3 (1.03) | -0.1 (0.90)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -0.3 (1.23) | -0.4 (1.06) | -0.2 (1.28)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | 0.0 (1.16) | 0.1 (1.06) | -0.2 (1.47)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | -0.2 (1.35) | -0.3 (1.40) | -0.1 (1.01)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -0.3 (1.12) | -0.1 (1.28) | -0.4 (1.30)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | 0.0 (1.83) | 0.3 (1.41) | -0.3 (1.51)

28. Secondary Outcome: Change From Baseline in Visual Analog Scale (Burning)
Description: Participants rated ocular symptom of burning by placing a vertical mark on the horizontal line to indicate the level of discomfort. 0 mm corresponds to "no discomfort" and 100 mm corresponds to "maximal discomfort."
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
mm
  Day 1 Pre-CAE | 30.4 (28.53) | 29.3 (26.74) | 22.4 (24.60)
  Day 1 Post-CAE: number analyzed (Participants) | 50 | 49 | 50
  Day 1 Post-CAE | 44.6 (29.99) | 44.1 (33.91) | 40.1 (32.15)
  Day 1 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 49 | 50
  Day 1 (Change from Pre-CAE to Post-CAE) | 14.2 (23.57) | 14.5 (22.27) | 17.7 (22.75)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | -1.9 (19.34) | -4.5 (25.73) | 0.5 (16.66)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | -3.0 (19.75) | -6.7 (24.08) | 0.3 (11.84)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Post-CAE) | -1.6 (23.56) | -10.8 (24.27) | -2.2 (16.90)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | 1.4 (26.91) | -3.5 (21.46) | -2.6 (17.42)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 29 (Pre-CAE) | -3.0 (26.13) | -6.6 (26.82) | -0.4 (15.67)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -7.3 (21.43) | -8.8 (26.93) | -3.2 (16.00)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -0.2 (23.76) | 2.4 (25.72) | -4.0 (24.77)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | -3.5 (27.19) | -10.0 (31.76) | -1.5 (16.19)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -1.3 (20.26) | -10.3 (26.98) | -4.6 (21.47)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | 2.2 (33.08) | 2.2 (30.19) | -3.0 (23.35)

29. Secondary Outcome: Change From Baseline in Visual Analog Scale (Itching)
Description: Participants rated ocular symptom of itching by placing a vertical mark on the horizontal line to indicate the level of discomfort. 0 mm corresponds to "no discomfort" and 100 mm corresponds to "maximal discomfort."
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
mm
  Day 1 Pre-CAE | 28.6 (27.09) | 26.2 (29.26) | 26.8 (23.70)
  Day 1 Post-CAE: number analyzed (Participants) | 50 | 49 | 50
  Day 1 Post-CAE | 37.0 (30.45) | 31.9 (33.26) | 35.0 (28.92)
  Day 1 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 49 | 50
  Day 1 (Change from Pre-CAE to Post-CAE) | 8.4 (21.67) | 5.2 (18.00) | 8.2 (22.76)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | -6.0 (19.05) | -2.8 (22.23) | 0.5 (19.54)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | -3.1 (19.18) | -4.5 (18.28) | 1.6 (20.27)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Post-CAE) | -8.0 (22.37) | -2.4 (19.21) | 1.9 (16.56)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -4.9 (27.23) | 2.2 (21.18) | 0.3 (19.52)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 29 (Pre-CAE) | -2.7 (24.78) | -9.5 (20.74) | -1.7 (20.97)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -9.3 (19.47) | -6.2 (23.64) | 2.2 (23.30)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -3.6 (15.78) | 5.2 (26.67) | 3.6 (25.99)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | -6.8 (22.73) | -8.1 (27.02) | -1.2 (23.65)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -7.0 (27.35) | -5.7 (23.95) | -2.1 (19.13)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -0.2 (25.65) | 4.7 (22.75) | 0.2 (26.94)

30. Secondary Outcome: Change From Baseline in Visual Analog Scale (Foreign Body)
Description: Participants rated ocular symptom of foreign body by placing a vertical mark on the horizontal line to indicate the level of discomfort. 0 mm corresponds to "no discomfort" and 100 mm corresponds to "maximal discomfort."
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
mm
  Day 1 Pre-CAE | 35.3 (25.95) | 35.1 (29.19) | 34.1 (25.87)
  Day 1 Post-CAE: number analyzed (Participants) | 50 | 49 | 50
  Day 1 Post-CAE | 45.1 (29.54) | 43.1 (31.03) | 49.9 (27.82)
  Day 1 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 49 | 50
  Day 1 (Change from Pre-CAE to Post-CAE) | 9.8 (24.25) | 8.1 (22.30) | 15.8 (21.57)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | -6.2 (23.33) | -3.4 (16.32) | -0.4 (19.69)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | -7.8 (23.00) | -1.3 (18.83) | -5.0 (17.15)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Post-CAE) | -8.5 (20.45) | -0.7 (21.90) | -7.9 (18.96)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -0.6 (28.16) | 0.8 (27.76) | -2.8 (20.72)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 29 (Pre-CAE) | -6.2 (28.69) | -5.0 (16.97) | -5.9 (26.37)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -8.6 (16.41) | -4.7 (19.58) | -1.1 (20.54)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | 1.4 (19.18) | 2.6 (19.77) | -0.6 (22.53)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | -9.3 (21.64) | -7.3 (28.49) | -5.2 (18.58)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -10.3 (23.81) | -1.5 (27.06) | -8.5 (19.20)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -1.0 (27.77) | 6.9 (30.44) | -3.7 (25.32)

31. Secondary Outcome: Change From Baseline in Visual Analog Scale (Blurred Vision)
Description: Participants rated ocular symptom of blurred vision by placing a vertical mark on the horizontal line to indicate the level of discomfort. 0 mm corresponds to "no discomfort" and 100 mm corresponds to "maximal discomfort."
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
mm
  Day 1 Pre-CAE | 18.5 (22.85) | 24.0 (27.00) | 26.9 (20.32)
  Day 1 Post-CAE: number analyzed (Participants) | 50 | 49 | 50
  Day 1 Post-CAE | 26.4 (28.30) | 32.2 (30.82) | 41.1 (28.62)
  Day 1 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 49 | 50
  Day 1 (Change from Pre-CAE to Post-CAE) | 7.9 (18.33) | 8.2 (25.15) | 14.2 (20.98)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | 2.5 (12.34) | -4.5 (23.77) | -4.2 (15.37)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | 3.7 (11.94) | -2.9 (19.40) | -2.1 (15.80)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Post-CAE) | -1.1 (14.37) | -7.3 (24.44) | -8.7 (21.87)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -4.7 (16.88) | -4.4 (23.96) | -6.6 (27.55)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 29 (Pre-CAE) | -2.0 (14.81) | -4.0 (18.45) | -3.2 (16.29)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -5.9 (16.34) | -7.9 (23.39) | -6.1 (17.73)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -2.5 (19.24) | -5.4 (21.62) | -7.7 (21.60)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | 0.5 (14.90) | -3.0 (21.79) | -1.2 (19.67)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -4.0 (19.15) | -6.9 (24.83) | -7.8 (21.29)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -4.5 (17.82) | -3.3 (27.89) | -6.5 (27.14)

32. Secondary Outcome: Change From Baseline in Visual Analog Scale (Dryness)
Description: Participants rated ocular symptom of dryness by placing a vertical mark on the horizontal line to indicate the level of discomfort. 0 mm corresponds to "no discomfort" and 100 mm corresponds to "maximal discomfort."
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
mm
  Day 1 Pre-CAE | 57.7 (20.98) | 58.6 (24.58) | 58.0 (22.90)
  Day 1 Post-CAE: number analyzed (Participants) | 50 | 49 | 50
  Day 1 Post-CAE | 74.2 (18.66) | 71.8 (21.47) | 75.0 (18.09)
  Day 1 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 49 | 50
  Day 1 (Change from Pre-CAE to Post-CAE) | 16.5 (16.76) | 13.3 (17.80) | 17.0 (18.30)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | -4.7 (16.31) | -2.1 (14.26) | -1.6 (19.15)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | -6.7 (19.32) | -7.4 (17.94) | -4.2 (20.52)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Post-CAE) | -1.7 (12.82) | -4.5 (16.69) | -1.7 (17.81)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | 5.0 (21.30) | 3.0 (21.22) | 2.5 (22.67)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 29 (Pre-CAE) | -6.4 (23.40) | -10.3 (19.89) | -7.1 (25.61)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -5.8 (14.15) | -7.1 (13.36) | -5.1 (12.50)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | 2.3 (21.34) | 3.5 (20.86) | 0.6 (23.70)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | -11.7 (24.14) | -11.3 (26.02) | -8.4 (26.81)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -8.3 (15.28) | -3.8 (14.57) | -7.7 (22.21)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | 3.3 (25.71) | 9.0 (24.83) | 1.7 (25.52)

33. Secondary Outcome: Change From Baseline in Visual Analog Scale (Photophobia)
Description: Participants rated ocular symptom of photophobia by placing a vertical mark on the horizontal line to indicate the level of discomfort. 0 mm corresponds to "no discomfort" and 100 mm corresponds to "maximal discomfort."
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
mm
  Day 1 Pre-CAE | 32.8 (28.41) | 37.4 (33.86) | 36.7 (29.19)
  Day 1 Post-CAE: number analyzed (Participants) | 50 | 49 | 50
  Day 1 Post-CAE | 38.1 (29.80) | 39.8 (34.50) | 49.7 (32.33)
  Day 1 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 49 | 50
  Day 1 (Change from Pre-CAE to Post-CAE) | 5.3 (16.70) | 2.2 (21.20) | 13.0 (22.01)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | 1.4 (16.17) | -5.0 (21.40) | -2.7 (18.46)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | -1.4 (16.19) | -11.0 (22.36) | -2.1 (18.17)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Post-CAE) | -2.4 (14.21) | -5.7 (19.94) | -8.8 (18.47)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -1.0 (19.59) | 5.8 (23.32) | -6.7 (22.12)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 29 (Pre-CAE) | -3.1 (19.61) | -7.3 (28.18) | -3.1 (26.01)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -4.0 (13.84) | -4.9 (18.11) | -0.9 (18.18)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | 3.0 (17.38) | 2.1 (13.89) | -2.7 (27.46)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | -4.1 (20.87) | -3.6 (26.95) | -3.6 (22.33)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -4.0 (21.66) | -2.3 (20.85) | -10.4 (23.91)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | 0.2 (28.34) | 1.5 (21.40) | -6.5 (24.53)

34. Secondary Outcome: Change From Baseline in Visual Analog Scale (Pain)
Description: Participants rated ocular symptom of pain by placing a vertical mark on the horizontal line to indicate the level of discomfort. 0 mm corresponds to "no discomfort" and 100 mm corresponds to "maximal discomfort."
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
mm
  Day 1 Pre-CAE | 17.0 (22.31) | 17.8 (23.62) | 17.4 (21.01)
  Day 1 Post-CAE: number analyzed (Participants) | 50 | 49 | 50
  Day 1 Post-CAE | 29.1 (30.50) | 26.3 (29.53) | 27.1 (29.83)
  Day 1 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 49 | 50
  Day 1 (Change from Pre-CAE to Post-CAE) | 12.1 (19.65) | 8.3 (15.81) | 9.7 (20.73)
  Change from Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change from Baseline: Day 8 | -2.2 (11.94) | -1.8 (22.41) | -2.6 (13.91)
  Change from Baseline: Day 15 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Pre-CAE) | 1.8 (20.34) | -3.1 (22.90) | -2.1 (14.54)
  Change from Baseline: Day 15 (Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 15 (Post-CAE) | -3.9 (17.59) | -2.0 (16.84) | -2.8 (18.66)
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from baseline: Day 15 (Change from Pre-CAE to Post-CAE) | -5.7 (19.81) | 1.5 (22.96) | -0.8 (23.07)
  Change from Baseline: Day 29 (Pre-CAE): number analyzed (Participants) | 50 | 48 | 50
  Change from Baseline: Day 29 (Pre-CAE) | -3.8 (17.30) | -3.3 (20.23) | -3.4 (15.35)
  Change from Baseline: Day 29 (Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from Baseline: Day 29 (Post-CAE) | -8.0 (16.05) | -1.8 (18.57) | -9.9 (18.61)
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 29 | 26 | 28
  Change from baseline: Day 29 (Change from Pre-CAE to Post-CAE) | -3.3 (15.38) | 7.7 (16.05) | -8.1 (20.05)
  Change from Baseline: Day 57 (Pre-CAE): number analyzed (Participants) | 46 | 44 | 50
  Change from Baseline: Day 57 (Pre-CAE) | -0.2 (22.85) | -6.6 (24.80) | -2.8 (14.32)
  Change from Baseline: Day 57 (Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from Baseline: Day 57 (Post-CAE) | -10.9 (16.16) | -4.1 (20.22) | -2.1 (12.68)
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE): number analyzed (Participants) | 46 | 43 | 49
  Change from baseline: Day 57 (Change from Pre-CAE to Post-CAE) | -10.7 (28.15) | 3.9 (21.67) | 0.7 (16.52)

35. Secondary Outcome: Change From Baseline in Ocular Surface and Disease Index (OSDI©)
Description: The OSDI is a simple 12-question survey that rates the severity of the participant's dry eye disease based on the symptoms. It is assessed on a scale of 0 to 100, with higher score representing greater disability.
Time Frame: Baseline (Day 1); Days 8, 15, 29, and 57
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
score on a scale
  Day 1 | 32.45 (14.379) | 36.78 (18.209) | 38.08 (16.602)
  Change From Baseline: Day 8: number analyzed (Participants) | 50 | 48 | 49
  Change From Baseline: Day 8 | -1.57 (7.885) | -0.87 (7.889) | -3.79 (8.161)
  Change From Baseline: Day 15: number analyzed (Participants) | 50 | 48 | 50
  Change From Baseline: Day 15 | -0.49 (9.048) | -2.98 (10.361) | -3.65 (10.727)
  Change From Baseline: Day 29: number analyzed (Participants) | 50 | 48 | 50
  Change From Baseline: Day 29 | -0.92 (10.324) | -4.42 (12.540) | -5.48 (12.471)
  Change From Baseline: Day 57: number analyzed (Participants) | 46 | 44 | 50
  Change From Baseline: Day 57 | -1.45 (11.598) | -3.33 (11.978) | -5.05 (10.817)

36. Secondary Outcome: Ora Calibra® Drop Comfort Scale
Description: Ora Calibra® drop comfort scale ranges from 0 to 10. A score of 0 indicates comfortable and 10 indicates uncomfortable. Lower score indicated better comfort level.
Time Frame: Upon instillation and 1 and 2 minutes post-instillation on Day 1
Population: The ITT Population with available data. The analysis was carried out with observed data only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 50 | 50 | 50
score on a scale
  Upon instillation on Day 1 | 2.8 (2.25) | 3.6 (2.40) | 3.3 (2.69)
  1 minute post-instillation on Day 1 | 2.0 (1.86) | 2.6 (1.93) | 2.3 (1.84)
  2 minutes post-instillation on Day 1 | 1.6 (1.75) | 2.3 (1.91) | 2.0 (1.89)

37. Secondary Outcome: Daily Diary: Change From Baseline in Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire for Dry Eye (Overall Ocular Discomfort)
Description: Ora Calibra® ocular discomfort & 4-symptom questionnaire for dry eye includes rating of the severity of 5 symptoms: ocular discomfort, burning, dryness, grittiness, and stinging.
  Participants rated the severity of overall ocular discomfort twice a day in a diary on 0 to 5 scale, where 0=none and 5=severe. Higher score represent higher severity.
  The average of the morning and evening assessments were calculated for each day. Weekly average scores were calculated based on the daily scores in the week.
Time Frame: From Baseline (Day 1) to Day 56
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 47 | 50 | 49
score on a scale
  Baseline: Daily average | 2.74 (0.884) | 2.82 (0.934) | 2.66 (0.789)
  Average Day 1 to Day 7: Change from Baseline Daily Average | -0.13 (0.326) | -0.09 (0.337) | -0.07 (0.376)
  Average Day 8 to Day 14: Change from Baseline Daily Average | -0.24 (0.430) | -0.10 (0.442) | -0.09 (0.510)
  Average Day 15 to Day 21: Change from Baseline Daily Average: number analyzed (Participants) | 47 | 48 | 49
  Average Day 15 to Day 21: Change from Baseline Daily Average | -0.21 (0.534) | -0.19 (0.465) | -0.13 (0.628)
  Average Day 22 to Day 28: Change from Baseline Daily Average: number analyzed (Participants) | 47 | 48 | 49
  Average Day 22 to Day 28: Change from Baseline Daily Average | -0.23 (0.558) | -0.29 (0.464) | -0.24 (0.650)
  Average Day 29 to Day 35: Change from Baseline Daily Average: number analyzed (Participants) | 47 | 48 | 48
  Average Day 29 to Day 35: Change from Baseline Daily Average | -0.18 (0.600) | -0.25 (0.548) | -0.15 (0.623)
  Average Day 36 to Day 42: Change from Baseline Daily Average: number analyzed (Participants) | 44 | 47 | 48
  Average Day 36 to Day 42: Change from Baseline Daily Average | -0.28 (0.597) | -0.28 (0.638) | -0.18 (0.638)
  Average Day 43 to Day 49: Change from Baseline Daily Average: number analyzed (Participants) | 44 | 46 | 48
  Average Day 43 to Day 49: Change from Baseline Daily Average | -0.34 (0.636) | -0.31 (0.666) | -0.16 (0.662)
  Average Day 50 to Day 56: Change from Baseline Daily Average: number analyzed (Participants) | 43 | 46 | 48
  Average Day 50 to Day 56: Change from Baseline Daily Average | -0.38 (0.713) | -0.29 (0.658) | -0.16 (0.674)

38. Secondary Outcome: Daily Diary: Change From Baseline in Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire for Dry Eye (Burning)
Description: Ora Calibra® ocular discomfort & 4-symptom questionnaire for dry eye includes rating of the severity of 5 symptoms: ocular discomfort, burning, dryness, grittiness, and stinging.
  Participants rated the severity of burning twice a day in a diary on 0 to 5 scale, where 0=none and 5=severe. Higher score represent higher severity.
  The average of the morning and evening assessments were calculated for each day. Weekly average scores were calculated based on the daily scores in the week.
Time Frame: From Baseline (Day 1) to Day 56
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 49 | 50 | 50
score on a scale
  Baseline: Daily average | 1.72 (1.126) | 1.49 (1.134) | 1.50 (1.135)
  Average Day 1 to Day 7: Change from Baseline Daily Average | -0.13 (0.309) | -0.08 (0.398) | -0.07 (0.328)
  Average Day 8 to Day 14: Change from Baseline Daily Average | -0.26 (0.369) | -0.17 (0.438) | -0.11 (0.420)
  Average Day 15 to Day 21: Change from Baseline Daily Average: number analyzed (Participants) | 49 | 48 | 50
  Average Day 15 to Day 21: Change from Baseline Daily Average | -0.22 (0.430) | -0.21 (0.498) | -0.12 (0.464)
  Average Day 22 to Day 28: Change from Baseline Daily Average: number analyzed (Participants) | 49 | 48 | 50
  Average Day 22 to Day 28: Change from Baseline Daily Average | -0.26 (0.449) | -0.29 (0.511) | -0.18 (0.546)
  Average Day 29 to Day 35: Change from Baseline Daily Average: number analyzed (Participants) | 49 | 48 | 49
  Average Day 29 to Day 35: Change from Baseline Daily Average | -0.18 (0.506) | -0.28 (0.523) | -0.11 (0.511)
  Average Day 36 to Day 42: Change from Baseline Daily Average: number analyzed (Participants) | 46 | 47 | 49
  Average Day 36 to Day 42: Change from Baseline Daily Average | -0.25 (0.440) | -0.35 (0.701) | -0.17 (0.500)
  Average Day 43 to Day 49: Change from Baseline Daily Average: number analyzed (Participants) | 46 | 46 | 49
  Average Day 43 to Day 49: Change from Baseline Daily Average | -0.25 (0.565) | -0.33 (0.647) | -0.13 (0.564)
  Average Day 50 to Day 56: Change from Baseline Daily Average: number analyzed (Participants) | 45 | 46 | 49
  Average Day 50 to Day 56: Change from Baseline Daily Average | -0.27 (0.571) | -0.33 (0.739) | -0.11 (0.527)

39. Secondary Outcome: Daily Diary: Change From Baseline in Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire for Dry Eye (Dryness)
Description: Ora Calibra® ocular discomfort & 4-symptom questionnaire for dry eye includes rating of the severity of 5 symptoms: ocular discomfort, burning, dryness, grittiness, and stinging.
  Participants rated the severity of dryness twice a day in a diary on 0 to 5 scale, where 0=none and 5=severe. Higher score represent higher severity.
  The average of the morning and evening assessments were calculated for each day. Weekly average scores were calculated based on the daily scores in the week.
Time Frame: From Baseline (Day 1) to Day 56
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 49 | 50 | 50
score on a scale
  Baseline: Daily average | 2.88 (0.793) | 2.96 (0.968) | 2.99 (0.669)
  Average Day 1 to Day 7: Change from Baseline Daily Average | -0.13 (0.391) | -0.11 (0.275) | -0.10 (0.383)
  Average Day 8 to Day 14: Change from Baseline Daily Average | -0.20 (0.505) | -0.14 (0.388) | -0.13 (0.504)
  Average Day 15 to Day 21: Change from Baseline Daily Average: number analyzed (Participants) | 49 | 48 | 50
  Average Day 15 to Day 21: Change from Baseline Daily Average | -0.20 (0.615) | -0.25 (0.479) | -0.13 (0.621)
  Average Day 22 to Day 28: Change from Baseline Daily Average: number analyzed (Participants) | 49 | 48 | 50
  Average Day 22 to Day 28: Change from Baseline Daily Average | -0.23 (0.620) | -0.30 (0.519) | -0.29 (0.659)
  Average Day 29 to Day 35: Change from Baseline Daily Average: number analyzed (Participants) | 49 | 48 | 49
  Average Day 29 to Day 35: Change from Baseline Daily Average | -0.17 (0.691) | -0.29 (0.485) | -0.21 (0.690)
  Average Day 36 to Day 42: Change from Baseline Daily Average: number analyzed (Participants) | 46 | 47 | 49
  Average Day 36 to Day 42: Change from Baseline Daily Average | -0.30 (0.680) | -0.32 (0.628) | -0.23 (0.677)
  Average Day 43 to Day 49: Change from Baseline Daily Average: number analyzed (Participants) | 46 | 46 | 49
  Average Day 43 to Day 49: Change from Baseline Daily Average | -0.35 (0.728) | -0.31 (0.704) | -0.25 (0.768)
  Average Day 50 to Day 56: Change from Baseline Daily Average: number analyzed (Participants) | 45 | 46 | 49
  Average Day 50 to Day 56: Change from Baseline Daily Average | -0.40 (0.793) | -0.29 (0.703) | -0.27 (0.812)

40. Secondary Outcome: Daily Diary: Change From Baseline in Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire for Dry Eye (Grittiness)
Description: Ora Calibra® ocular discomfort & 4-symptom questionnaire for dry eye includes rating of the severity of 5 symptoms: ocular discomfort, burning, dryness, grittiness, and stinging.
  Participants rated the severity of grittiness twice a day in a diary on 0 to 5 scale, where 0=none and 5=severe. Higher score represent higher severity.
  The average of the morning and evening assessments were calculated for each day. Weekly average scores were calculated based on the daily scores in the week.
Time Frame: From Baseline (Day 1) to Day 56
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 49 | 50 | 50
score on a scale
  Baseline: Daily average | 2.14 (0.988) | 1.84 (1.248) | 2.07 (1.177)
  Average Day 1 to Day 7: Change from Baseline Daily Average | -0.19 (0.450) | -0.07 (0.331) | -0.03 (0.407)
  Average Day 8 to Day 14: Change from Baseline Daily Average | -0.27 (0.555) | -0.07 (0.500) | -0.08 (0.555)
  Average Day 15 to Day 21: Change from Baseline Daily Average: number analyzed (Participants) | 49 | 48 | 50
  Average Day 15 to Day 21: Change from Baseline Daily Average | -0.22 (0.594) | -0.16 (0.540) | -0.14 (0.554)
  Average Day 22 to Day 28: Change from Baseline Daily Average: number analyzed (Participants) | 49 | 48 | 50
  Average Day 22 to Day 28: Change from Baseline Daily Average | -0.26 (0.628) | -0.21 (0.615) | -0.23 (0.655)
  Average Day 29 to Day 35: Change from Baseline Daily Average: number analyzed (Participants) | 49 | 48 | 49
  Average Day 29 to Day 35: Change from Baseline Daily Average | -0.21 (0.724) | -0.22 (0.554) | -0.18 (0.627)
  Average Day 36 to Day 42: Change from Baseline Daily Average: number analyzed (Participants) | 46 | 47 | 49
  Average Day 36 to Day 42: Change from Baseline Daily Average | -0.35 (0.682) | -0.18 (0.642) | -0.18 (0.561)
  Average Day 43 to Day 49: Change from Baseline Daily Average: number analyzed (Participants) | 46 | 46 | 49
  Average Day 43 to Day 49: Change from Baseline Daily Average | -0.38 (0.682) | -0.16 (0.833) | -0.16 (0.666)
  Average Day 50 to Day 56: Change from Baseline Daily Average: number analyzed (Participants) | 45 | 46 | 49
  Average Day 50 to Day 56: Change from Baseline Daily Average | -0.36 (0.764) | -0.11 (0.959) | -0.18 (0.708)

41. Secondary Outcome: Daily Diary: Change From Baseline in Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire for Dry Eye (Stinging)
Description: Ora Calibra® ocular discomfort & 4-symptom questionnaire for dry eye includes rating of the severity of 5 symptoms: ocular discomfort, burning, dryness, grittiness, and stinging.
  Participants rated the severity of stinging twice a day in a diary on 0 to 5 scale, where 0=none and 5=severe. Higher score represent higher severity.
  The average of the morning and evening assessments were calculated for each day. Weekly average scores were calculated based on the daily scores in the week.
Time Frame: From Baseline (Day 1) to Day 56
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
Number analyzed (Participants) | 49 | 50 | 50
score on a scale
  Baseline: Daily average | 1.53 (1.113) | 1.20 (1.127) | 1.26 (1.075)
  Average Day 1 to Day 7: Change from Baseline Daily Average | -0.14 (0.349) | -0.13 (0.327) | -0.11 (0.342)
  Average Day 8 to Day 14: Change from Baseline Daily Average | -0.24 (0.409) | -0.12 (0.438) | -0.14 (0.469)
  Average Day 15 to Day 21: Change from Baseline Daily Average: number analyzed (Participants) | 49 | 48 | 50
  Average Day 15 to Day 21: Change from Baseline Daily Average | -0.16 (0.428) | -0.22 (0.515) | -0.20 (0.455)
  Average Day 22 to Day 28: Change from Baseline Daily Average: number analyzed (Participants) | 49 | 48 | 50
  Average Day 22 to Day 28: Change from Baseline Daily Average | -0.12 (0.517) | -0.28 (0.533) | -0.24 (0.546)
  Average Day 29 to Day 35: Change from Baseline Daily Average: number analyzed (Participants) | 49 | 48 | 49
  Average Day 29 to Day 35: Change from Baseline Daily Average | -0.11 (0.572) | -0.28 (0.538) | -0.21 (0.517)
  Average Day 36 to Day 42: Change from Baseline Daily Average: number analyzed (Participants) | 46 | 47 | 49
  Average Day 36 to Day 42: Change from Baseline Daily Average | -0.22 (0.564) | -0.32 (0.631) | -0.20 (0.514)
  Average Day 43 to Day 49: Change from Baseline Daily Average: number analyzed (Participants) | 46 | 46 | 49
  Average Day 43 to Day 49: Change from Baseline Daily Average | -0.24 (0.553) | -0.27 (0.647) | -0.16 (0.612)
  Average Day 50 to Day 56: Change from Baseline Daily Average: number analyzed (Participants) | 45 | 46 | 49
  Average Day 50 to Day 56: Change from Baseline Daily Average | -0.22 (0.575) | -0.28 (0.744) | -0.15 (0.577)

ADVERSE EVENTS:
Time Frame: Baseline up to 8 weeks
Description: Safety population included all randomized subjects who have received at least one dose of the investigational product.
Arm/Group | 0.10% HL036 Ophthalmic Solution | 0.25% HL036 Ophthalmic Solution | Placebo
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 13/50 | 13/50 | 9/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.10% HL036 Ophthalmic Solution (N=50) | 0.25% HL036 Ophthalmic Solution (N=50) | Placebo (N=50)
Conjunctivitis allergic (Eye disorders) | 3 | 4 | 0
Visual acuity reduced (Eye disorders) | 3 | 0 | 0
Instillation site pain (General disorders) | 2 | 6 | 1
Nasopharyngitis (Infections and infestations) | 5 | 3 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/39/NCT03334539/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT03334539/SAP_001.pdf